CLINICAL TRIAL: NCT00730223
Title: Genetic Determinants of the Metabolism of Non-nucleoside Reverse Transcriptase Inhibitors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, David Haas, Professor of Medicine, Vanderbilt University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 040062; GM31304; CFAR Discovery Grant
Record Dates: First submitted 2008-08-04; First posted 2008-08-08 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: HIV Infections
Keywords: Nevirapine; Efavirenz; pharmacokinetics; healthy; CYP2B6; HIV/AIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Nevirapine; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Nevirapine and Efavirenz — single oral dose 200mg of nevirapine and single oral dose 600 mg of efavirenz
  Other Names: Viramune; Sustiva

SUMMARY:
To see if certain variations in the CYP2B6 gene contribute to differences in plasma drug levels and central nervous system side affects in people who take nevirapine or efavirenz.

ELIGIBILITY:
Inclusion Criteria:

* Healthy African American men and women.
* 18-55 years of age.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Currently or recently (within the previous 30 days) received medications known or likely to be metabolized by, or interact wth the CYP450 enzymes.
* Prior or current hepatic or psychiatric disease illness that in the judgment of the investigator would interfere in the study performance.
* Active alcohol or illicit drug abuse use that in the judgment of the investigator would interfere in the study performance.
* Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) >1.5 X upper limit of normal.
* Positive pregnancy test in women of childbearing potential.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2004-03; Primary Completion 2006-03 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of single dose nevirapine and single dose efavirenz | 5-6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David W Haas, MD, Principal Investigator — Associate Professor of Medicine